CLINICAL TRIAL: NCT04533256
Title: Effects of Renal Replacement Therapy With Hemoadsoption in Patients With Sepsis
Status: Completed | Type: Observational
Sponsor: Institutul Clinic Fundeni (Other)
Responsible Party: Principal Investigator, Popescu Mihai, clinical professor, Institutul Clinic Fundeni
Other Study IDs: Cyto-Sepsis
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Sepsis
Keywords: organ failure; renal replacement therapy; hemoadsorption
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Procedure: CytoSorb — three consecutive sessions of hemoadsorption in patients with sepsis

SUMMARY:
Hemoadsorption has been demonstrated to improve clinical and paraclinical results in critically ill patients with sepsis and septic shock. The present study investigates the effects of three consecutive sessions of hemoadsorption, performed in accordance to the local protocol for treating patients with sepsis, on organ failure, severity scores and 30-days mortality. Paraclinical results and severity scores were obtained before and after the three consecutive sessions.

ELIGIBILITY:
Inclusion Criteria:

* patients with sepsis or septic shock who require hemoadsorption in accordance with local guidelines

Exclusion Criteria:

* unsigned informed consent
* duration of therapy under 12 hours
* death before the three consecutive sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sepsis or septic shock who require hemoadsorption in accordance with local guidelines. The decision of hemoadsorption is made by the attending physician prior to study inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-07-10 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
28-days mortality | 28 days after ICU admission
  28-days mortality

SECONDARY OUTCOMES:
severity score | 3 days
  dynamics of SOFA score (Sequential Organ Failure Assessment) calculated as the mathematical difference in post-therapy SOFA score and pre-therapy SOFA score

CONTACTS AND LOCATIONS:
Overall Officials: Dana Tomescu, Prof, Study Chair — Fundeni Clinical Institute
Locations (1):
- Fundeni Clinical Institute, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: Undecided